CLINICAL TRIAL: NCT02233790
Title: Comparison of Ticagrelor and Clopidogrel on Reperfusion in Patients With AMI Undergoing PPCI Evaluated by SPECT
Brief Title: Ticagrelor and Clopidogrel on Reperfusion in Patients With AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Hospital of China Medical University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Yingxian Sun, Director, Department of cardiology, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0209
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Infarction; No-Reflow Phenomenon
Keywords: Myocardial infarction; No-Reflow Phenomenon; Ticagrelor; Clopidogrel; Single-Photon Emission Computerized Tomography
MeSH Terms: conditions — Myocardial Infarction; No-Reflow Phenomenon | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — a loading dose of 180mg pre-PCI, and then 90 mg twice daily for 1 Month within the study. Thereafter, the patients will take clopidogrel if Ticagrelor is not available on the market.
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Clopidogrel — Clopidogrel 75 mg once daily after a loading dose of 300 mg pre-PCI.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The patients with acute myocardial infarction (AMI) present high mortality and morbidity rate,even treated with stenting in the blocked heart vessels.

The appearance of no-reflow is common after re-opening of the blocked vessel. The no-reflow were commonly attributed to tiny blockage in coronary micro-vasculature by thrombus and spasm of the micro-vessel during stenting.

An agent with more effective anti-clotting and micro-vessel dilation would be helpful to solve the issue of no-reflow. Ticagrelor was demonstrated to be a potent platelet inhibitor and a potent micro-vessel dilator which can influence metabolism of adenosine, a endogenous potent small vessel dilator.

This study is to test the effectiveness of ticagrelor on improving reperfusion and minimizing the myocardial infarct size after PPCI in patients with AMI.

DETAILED DESCRIPTION:
The patients with acute myocardial infarction (AMI) present high mortality and morbidity rate, and also have malignant prognosis even if they could survive. The mortality and prognosis has been improved markedly because of the treatment with primary percutaneous coronary intervention (PPCI). However, the issue of no-reflow after revascularization has not been solved yet. The mechanisms of no-reflow in human being were regarded mainly as micro-embolism in coronary micro-circulation with thrombus or debris from atherosclerotic plaque, coronary micro-vasculature spasm and other conditions.

Therefore, an agent with potent antithrombotic and micro-vasculature dilation function would be more effective on prevention of no-reflow after coronary revascularization. Ticagrelor was demonstrated to be a potent platelet inhibitor and a potent micro-vessel dilator which can influence metabolism of adenosine.

Ticagrelor can inhibit adenosine uptake in vitro and subsequently augments cardiac blood flow in a canine model of reactive hypoxia- or adenosine-induced blood flow increases. In a dog coronary thrombosis model, ticagrelor blocks ADP-induced platelet activation and aggregation; prevents platelet-mediated thrombosis; prolongs reperfusion time and reduces re-occlusion and cyclic flow variation; and significantly decreases infarct size and rapidly restores myocardial tissue perfusion. These findings suggest that ticagrelor may have additional benefits in patients with acute coronary syndrome beyond inhibition of platelet aggregation, which is advantageous to the dilation of microcirculation and improvement of myocardial perfusion. AMISTAD study shows that: adenosine reperfusion therapy can reduce 33% of the infarction area assessed by single-photon emission computed tomography (SPECT) detection. AMISTAD- 2 study showed that: adenosine early reperfusion therapy can reduce the composite end point of death and heart failure events. Additionally, ticagrelor is a non-precursor agent, playing a role directly on platelet inhibition.

Myocardial perfusion imaging with SPECT is among the most widely used and well-established noninvasive tools for the diagnosis of ischemic coronary disease. It has been shown to have a high sensitivity and specificity in identifying patients with coronary artery disease and to be accurate in identifying areas of prior myocardial infarction.

Given the evidence (from PLATO trial) of greater IPA with ticagrelor than clopidogrel, similar risk of major bleeding and probable effect of micro-vasculature dilation due to adenosine, ticagrelor will improve the reperfusion and decrease the infarct size significantly.

This study is to test the effectiveness of ticagrelor on improving reperfusion and minimizing the myocardial infarct size after PPCI in patients with AMI. Also, it is to evaluate the safety of ticagrelor in patients with AMI.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Patients with acute ST-segment elevation myocardial infarction, an onset of symptoms presented within 12 hours. Two criteria have to be met: persistent ST-segment elevation of at least 0.1 mV in at least two contiguous leads or a new left bundle-branch block, and the intention to perform primary PCI
* Patients must agree to undergo all protocol-required follow-up examinations and not to participate any other clinical trials within the duration of this study

Exclusion Criteria:

* Any contraindication against the use of clopidogrel or ticagrelor
* Fibrinolytic therapy within 24 hours before randomization
* Stroke within the previous 6 months or intracranial hemorrhage at any time before randomization
* Any other concomitant severe organic or systemic disorder, such as severe liver (ALT>3×ULN )or renal disease(creatinin>5.0mg/dl or 442μmol/L), etc.
* A need for oral anticoagulation therapy
* An increased risk of bradycardia or atrial-ventricle block
* Concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer
* Pregnant women or breast-feeding, or planning to become pregnant while enrolled in this study
* Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
myocardial infarcted size | 1 week
  To evaluate the infarcted size on Day 7 after PPCI by SPECT.

SECONDARY OUTCOMES:
elevated ST segment resolution | 1 hour and 24 hours
  To observe the elevated ST segment resolution at 1 h and 24 h after PPCI;

OTHER OUTCOMES:
severe brachycardia arrhythmia | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Yingxian Sun, Dr., Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Background] Mahaffey KW, Puma JA, Barbagelata NA, DiCarli MF, Leesar MA, Browne KF, Eisenberg PR, Bolli R, Casas AC, Molina-Viamonte V, Orlandi C, Blevins R, Gibbons RJ, Califf RM, Granger CB. Adenosine as an adjunct to thrombolytic therapy for acute myocardial infarction: results of a multicenter, randomized, placebo-controlled trial: the Acute Myocardial Infarction STudy of ADenosine (AMISTAD) trial. J Am Coll Cardiol. 1999 Nov 15;34(6):1711-20. doi: 10.1016/s0735-1097(99)00418-0. PMID 10577561
- [Background] Steg PG, James S, Harrington RA, Ardissino D, Becker RC, Cannon CP, Emanuelsson H, Finkelstein A, Husted S, Katus H, Kilhamn J, Olofsson S, Storey RF, Weaver WD, Wallentin L; PLATO Study Group. Ticagrelor versus clopidogrel in patients with ST-elevation acute coronary syndromes intended for reperfusion with primary percutaneous coronary intervention: A Platelet Inhibition and Patient Outcomes (PLATO) trial subgroup analysis. Circulation. 2010 Nov 23;122(21):2131-41. doi: 10.1161/CIRCULATIONAHA.109.927582. Epub 2010 Nov 8. PMID 21060072
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Ross AM, Gibbons RJ, Stone GW, Kloner RA, Alexander RW; AMISTAD-II Investigators. A randomized, double-blinded, placebo-controlled multicenter trial of adenosine as an adjunct to reperfusion in the treatment of acute myocardial infarction (AMISTAD-II). J Am Coll Cardiol. 2005 Jun 7;45(11):1775-80. doi: 10.1016/j.jacc.2005.02.061. PMID 15936605